CLINICAL TRIAL: NCT05536700
Title: Clinical Utility of Mass Spectrometry (EasyM) for Detecting Minimal Residual Disease (MRD) by Monitoring Serum Monoclonal Immunoglobulins in Multiple Myeloma
Brief Title: Using Mass Spectrometry (EasyM) Detecting Minimal Residual Disease (MRD) in Multiple Myeloma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Shanghai Kuaixu Biotechnology Co., Ltd (Unknown)
Responsible Party: Principal Investigator, AnGang,MD, Professor, Institute of Hematology & Blood Diseases Hospital, China
Other Study IDs: EasyM-MM-2021
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Multiple Myeloma
Keywords: mass spectrometry; serum immunoglobulin; minimal residual disease; MRD; EasyM; M protein
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The presence of minimal residual disease (MRD) is an important prognostic factor for multiple myeloma, while M-protein is a widely accepted biomarker used for multiple myeloma (MM) diagnose. Detecting MRD by monitoring M-protein using mass spectrometry (MS) is promising due to its high analytical sensitivity. To evaluate the correlation between MS-MRD and overall disease burden, over 60 patients with 500+ samples were identified for this study. The M-protein sequence and the patient-specific M-protein peptides of each patient were obtained by de novo protein sequencing platform using the diagnostic serum (> 30g/L). The follow- up samples were then measured by a parallel reaction monitoring (PRM) assay.

ELIGIBILITY:
Inclusion Criteria:

Subjects with available baseline and sequential serum samples.

Exclusion Criteria:

Subjects without baseline and sequential serum samples.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects diagnosed with MM.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Estimated)
Dates: Start 2021-12-31 (Actual); Primary Completion 2022-09-17 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Quantitative measurement of M protein | From June 6, 2022 to December 31, 2022
  Detecting the M protein concentration and its dynamic change curve

SECONDARY OUTCOMES:
sequence detection of M protein | From December 31, 2021 to May 31, 2022
  Detecting the M protein sequence in each person

CONTACTS AND LOCATIONS:
Overall Officials: InstituteHBDH, Principal Investigator — Institute of Hematology and Blood Diseases Hospital,Tianjin, China, 300020
Locations (1):
- InsituteHBDH, Tianjin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan H, Wang B, Shi L, Pan N, Yan W, Xu J, Gong L, Li L, Liu Y, Du C, Cui J, Zhu G, Deng S, Sui W, Xu Y, Yi S, Hao M, Zou D, Chen X, Qiu L, An G. Monitoring Minimal Residual Disease in Patients with Multiple Myeloma by Targeted Tracking Serum M-Protein Using Mass Spectrometry (EasyM). Clin Cancer Res. 2024 Mar 15;30(6):1131-1142. doi: 10.1158/1078-0432.CCR-23-2767. PMID 38170583